CLINICAL TRIAL: NCT03090451
Title: Evaluating the Dynamics of Insulin and Non-insulin Mediated Effects on Glucose During Aerobic Exercise in Subjects With Type 1 Diabetes
Brief Title: Exercise Physiology Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Joseph El Youssef, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16761
Record Dates: First submitted 2017-03-07; First posted 2017-03-24 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia
Keywords: Insulin; Glucose Clamp; Glucose Tracer; Artificial Pancreas; Exercise; Aerobic
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two main arms: 1) moderate aerobic exercise, 2) intense aerobic exercise. In each arm, subjects will undergo three separate studies, i) at low insulin levels, ii) at medium insulin levels, and iii) at high insulin levels.
Masking Description: No masking for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate Aerobic Exercise (Experimental): Subjects will undergo moderate aerobic physical exercise (40-45% of VO2-max) on three separate days at i) low insulin levels, ii) medium insulin levels, and iii) high insulin levels.
  Interventions: Behavioral: Aerobic Exercise
- Intense Aerobic Exercise (Experimental): Subjects will undergo intense aerobic physical exercise (60-65% of VO2-max) on three separate days at i) low insulin levels, ii) medium insulin levels, and iii) high insulin levels.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Aerobic physical exercise on treadmill, with intensity based on prior VO2-max testing during the screening visit.

SUMMARY:
People with type 1 diabetes often find exercise very difficult to manage, because of the high risk for low blood glucose levels. This can occur very quickly once exercise starts and presents many risks for subjects, such as severe symptoms, confusion, passing out, seizures, and even coma or death in very severe cases. Preventing low blood glucose levels during and after exercise is important because physical exercise is a key component of managing diabetes. It is often hard to correctly adjust insulin infusion rates or doses before exercise as the relationship between exercise and changes in glucose levels in those who have type 1 diabetes is still not fully understood. Therefore, the investigators propose this study to further our understanding in this area.

This study is designed to help separate the effects of insulin from those of muscle work (non-insulin effects) on the changes in blood glucose levels during aerobic exercise. The main hypothesis is that the non-insulin effects occur quickly during exercise and account for the rapid change in blood glucose levels once aerobic exercise begins. These effects can be separated from the slower changes in insulin sensitivity that occur because of exercise, and which account for reduced insulin demand even after exercise has stopped. The investigators will investigate the effects of both moderate and intense aerobic exercise at different levels of insulin in the body to help separate the insulin and non-insulin effects.

The investigators wish to recruit 26 subjects to take part in this study. Subjects will be randomly divided into two groups, with 13 in each group. Group 1 will undergo moderate aerobic exercise, while group 2 will undergo intense aerobic exercise. Each subject will repeat the exercise study three times on three separate days at least 2 weeks apart, while having insulin infused at a low, a medium, and a high rate. Subjects will have an IV line placed in each arm, one for drawing blood relatively frequently during the study, and another for infusion of insulin, glucose, and a special glucose tracer (non-radioactive). Each study lasts about 9 hours.

Information from this study will be used to help develop a mathematical model of how glucose changes during exercise in type 1 diabetes. Such a model of type 1 diabetes and exercise will be very useful for adjusting insulin doses in patients who use multiple daily injections of insulin, and can help to guide an automated insulin delivery system, such as the artificial pancreas.

DETAILED DESCRIPTION:
Diabetes mellitus afflicts close to 10% of our population and 5% of those with diabetes have type 1, which is defined by an absolute deficiency of insulin. The need for managing diabetes is critical, given the economic burden of this disease, with over $175 billion dollars in direct health care costs, and almost another $70 billion in indirect costs for disability and work loss. The personal impact is equally as important for people with this disease, as diabetes mellitus is the leading cause of blindness, the need for kidney dialysis, and non-traumatic amputations in the United States. Type 2 diabetes is associated with reduced insulin sensitivity and the metabolic syndrome, and dietary modification and exercise are important components in the management of underlying insulin resistance. However, these lifestyle strategies are also important in type 1 diabetes for many reasons: 1) type 1 diabetes subjects now live into adulthood, when insulin resistance and obesity become factors for glycemic control, 2) latent autoimmune diabetes of adulthood (LADA) represents a "mixed" form of autoimmune diabetes where some type 2 diabetes characteristics such as insulin resistance can exist, and 3) dietary modification and exercise remain effective means for management of acute hyperglycemia and, in the longer term, HbA1c, potentially reducing the risk of microvascular complications. Therefore, the need for exercise is still evident in subjects with type 1 diabetes to maintain good glycemic control and to prevent complications from developing. However, exercise is challenging for people with T1D to manage. Exercise causes increased insulin sensitivity along with rapid uptake of glucose by muscle and other tissues within the body, leading to a sharp decline in glucose levels and hypoglycemia as shown by other groups as well as ours.

Without adjustments in insulin for exercise, hypoglycemia is common in persons with type 1 diabetes. In a study of 48 individuals with T1D, with no adjustments to insulin, who exercise for 60 min at a moderate intensity, glucose levels dropped on average by 40%, with 52% of subjects falling to 70 mg/dL or below. Despite this clear need for insulin adjustments for exercise, there are no uniform recommendations on how to dose insulin around the time of exercise. In 2006, the DirecNet Study Group published a study on the impact of suspending basal insulin at the start of exercise in 40 children with type 1 diabetes on insulin pump therapy. This intervention significantly reduced hypoglycemia (from 43% to 16%), but much more commonly resulted in hyperglycemia (increased from 4% to 23%). Schiavon and Cobelli et al addressed this issue of how to best adjust insulin for exercise using in silico simulations. Adjusting insulin doses in the in silico environment decreased hypoglycemia from 88% to 16% of patients when a universal adjustment was applied, and to 4% when an individual adjustment was applied.

The study described within this protocol is designed to disambiguate the impact of exercise on insulin and non-insulin mediated effects on glycemic control. To achieve this, the investigators will perform a series of stable glucose tracer studies in which subjects will be fasting for about 8 hours and will undergo aerobic exercise at a moderate and intense level for 45 minutes while insulin rates are clamped at a low (subject's basal rate), medium (basal x 1.5), and high (basal x 3) insulin infusion rate. Subject's basal rates will be obtained from injected basal insulin amounts, such as NPH/glargine/detemir, or basal rates in those who use insulin pumps and will be adjusted for the HbA1c, as described in the OHSU AP system. Di-deuterated glucose (6,6-2H2-glucose) which is not radioactive and which can be metabolized via usual pathways in the human body will be the stable tracer. Each subject per arm will undergo 3 10-hour studies while blood glucose, insulin, and glucagon levels are captured throughout the study, and catecholamine and fatty acid levels are captured during and just after the exercise period, as outlined below. Glucose tracer levels will be measured at OHSU through the Bioanalytical Shared Resource/PK core lab, and calculation of rate of appearance (Ra) and rate of disappearance (Rd) of glucose will be performed by our colleagues at McGill University using a non-steady state model of glucose dynamics.

The data obtained from this study will inform an updated model of glucose regulation in type 1 diabetes, providing exercise as an input to the model, which will be utilized in a model predictive control (MPC) system for managing type 1 diabetes. Such a system can be used to deliver insulin and/or glucagon to manage glycemic changes during and outside of exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus for at least 1 year.
2. Male or female subjects 18 to 45 years of age.
3. Physically willing and able to perform 45 minutes of physical exercise, as determined by the investigator after reviewing the subject's activity level.
4. A hemoglobin A1c (HbA1c) less than 10%.
5. Willingness to follow all study procedures, including attending all study visits.
6. Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

1. Female of childbearing potential who is pregnant, intending to become pregnant, breast-feeding, or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill/patch/vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
2. Any cardiovascular disease, defined as clinically significant EKG abnormality at the time of screening, or any history of: stroke, heart failure, myocardial infarction, angina pectoris, coronary arterial bypass grafting, or angioplasty. Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia may be judged by the investigator to be exclusionary.
3. Renal insufficiency (GFR < 60 ml/min, using the MDRD equation as reported by the OHSU laboratory).
4. Liver failure, cirrhosis, or any other liver disease that compromises liver function as determined by the investigator.
5. Hematocrit of less than 34%.
6. Hypertension with systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg despite treatment or who have treatment-refractory hypertension (e.g. requiring four or more medications).
7. History of severe hypoglycemia during the past 12 months prior to screening visit or hypoglycemia unawareness as judged by the investigator. Subjects will complete a hypoglycemia awareness questionnaire (included in Appendix A). Subjects will be excluded for four or more 'R' responses.
8. Adrenal insufficiency.
9. Any active infection.
10. Known of suspected abuse of alcohol, narcotics, or illicit drugs.
11. Seizure disorder.
12. Active foot ulceration.
13. Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
14. Major surgical operation within 30 days prior to screening.
15. Use of an investigational drug within 30 days prior to screening.
16. Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
17. Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
18. Insulin resistance requiring more than 200 units per day.
19. Current administration of oral or parenteral corticosteroids.
20. Any life-threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal cell cancer of the skin).
21. Beta blockers or non-dihydropyridine calcium channel blockers.
22. Current use of any medication intended to lower glucose other than insulin (e.g. use of liraglutide, exenatide, etc.)
23. Diagnosis of pheochromocytoma, insulinoma, or glucagonoma, personal or family history of multiple endocrine neoplasia (MEN) 2A, MEN 2B, neurofibromatosis or von Hippel-Lindau disease.
24. History of severe hypersensitivity to milk protein.
25. Conditions that may result in low levels of releasable glucose in the liver and an inadequate reversal of hypoglycemia by glucagon such as prolonged fasting, starvation or chronic hypoglycemia as determined by the investigator.
26. A positive response to any of the questions from the Physical Activity Readiness Questionnaire with one exception: subject will not be excluded if only a single blood pressure medication that doesn't impact heart rate is used, and blood pressure is controlled on the medication (blood pressure is less than 140/90 mmHg). See Appendix B.
27. Any chest discomfort with physical activity, including pain or pressure, or other types of discomfort.
28. Any clinically significant disorder which, in the opinion of the investigator, may jeopardize the subject's safety or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Non-insulin mediated glucose uptake (NIMGU) | At baselin and at 30 minutes into physical exercise
  Rate of disappearance of glucose in [mg/kg]/min during exercise that is not related to the insulin effect, as calculated using a non-steady state model of glucose dynamics. This will be compared to the baseline NIMGU before exercise.

SECONDARY OUTCOMES:
Insulin mediated glucose uptake (IMGU) | At baseline and at 30 minutes into physical exercise
  Rate of disappearance of glucose in [mg/kg]/min during exercise that is related to the insulin effect, as calculated using a non-steady state model of glucose dynamics.This will be compared to the baseline IMGU before exercise.
Mean glucose level | 9 hours
  Mean glucose level throughout the study (without the run-in period)
Time spent in severe hypoglycemia | 9 hours
  Time in minutes spent in the range of glucose < 50 mg/dl.
Time spent in hypoglycemia | 9 hours
  Time in minutes spent in the range of glucose < 70 mg/dl.
Time spent in hyperglycemia | 9 hours
  Time in minutes spent in the range of glucose > 180 mg/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph El Youssef, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. in 2012. Diabetes Care. 2013 Apr;36(4):1033-46. doi: 10.2337/dc12-2625. Epub 2013 Mar 6. PMID 23468086
- [Background] Livingstone SJ, Levin D, Looker HC, Lindsay RS, Wild SH, Joss N, Leese G, Leslie P, McCrimmon RJ, Metcalfe W, McKnight JA, Morris AD, Pearson DW, Petrie JR, Philip S, Sattar NA, Traynor JP, Colhoun HM; Scottish Diabetes Research Network epidemiology group; Scottish Renal Registry. Estimated life expectancy in a Scottish cohort with type 1 diabetes, 2008-2010. JAMA. 2015 Jan 6;313(1):37-44. doi: 10.1001/jama.2014.16425. PMID 25562264
- [Background] Rusavy Z, Lacigova S. [Life expectancy of people with type 1 diabetes in the past and today]. Vnitr Lek. 2014 Sep;60(9):765-71. Czech. PMID 25294766
- [Background] Naik RG, Brooks-Worrell BM, Palmer JP. Latent autoimmune diabetes in adults. J Clin Endocrinol Metab. 2009 Dec;94(12):4635-44. doi: 10.1210/jc.2009-1120. Epub 2009 Oct 16. PMID 19837918
- [Background] Yardley JE, Hay J, Abou-Setta AM, Marks SD, McGavock J. A systematic review and meta-analysis of exercise interventions in adults with type 1 diabetes. Diabetes Res Clin Pract. 2014 Dec;106(3):393-400. doi: 10.1016/j.diabres.2014.09.038. Epub 2014 Oct 7. PMID 25451913
- [Background] Quirk H, Blake H, Tennyson R, Randell TL, Glazebrook C. Physical activity interventions in children and young people with Type 1 diabetes mellitus: a systematic review with meta-analysis. Diabet Med. 2014 Oct;31(10):1163-73. doi: 10.1111/dme.12531. PMID 24965376
- [Background] Breton MD, Brown SA, Karvetski CH, Kollar L, Topchyan KA, Anderson SM, Kovatchev BP. Adding heart rate signal to a control-to-range artificial pancreas system improves the protection against hypoglycemia during exercise in type 1 diabetes. Diabetes Technol Ther. 2014 Aug;16(8):506-11. doi: 10.1089/dia.2013.0333. Epub 2014 Apr 4. PMID 24702135
- [Background] Jacobs PG, Resalat N, El Youssef J, Reddy R, Branigan D, Preiser N, Condon J, Castle J. Incorporating an Exercise Detection, Grading, and Hormone Dosing Algorithm Into the Artificial Pancreas Using Accelerometry and Heart Rate. J Diabetes Sci Technol. 2015 Oct 5;9(6):1175-84. doi: 10.1177/1932296815609371. PMID 26438720
- [Background] Tansey MJ, Tsalikian E, Beck RW, Mauras N, Buckingham BA, Weinzimer SA, Janz KF, Kollman C, Xing D, Ruedy KJ, Steffes MW, Borland TM, Singh RJ, Tamborlane WV; Diabetes Research in Children Network (DirecNet) Study Group. The effects of aerobic exercise on glucose and counterregulatory hormone concentrations in children with type 1 diabetes. Diabetes Care. 2006 Jan;29(1):20-5. doi: 10.2337/diacare.29.1.20. PMID 16373890
- [Background] Diabetes Research in Children Network (DirecNet) Study Group; Tsalikian E, Kollman C, Tamborlane WB, Beck RW, Fiallo-Scharer R, Fox L, Janz KF, Ruedy KJ, Wilson D, Xing D, Weinzimer SA. Prevention of hypoglycemia during exercise in children with type 1 diabetes by suspending basal insulin. Diabetes Care. 2006 Oct;29(10):2200-4. doi: 10.2337/dc06-0495. PMID 17003293
- [Background] Schiavon M, Dalla Man C, Kudva YC, Basu A, Cobelli C. In silico optimization of basal insulin infusion rate during exercise: implication for artificial pancreas. J Diabetes Sci Technol. 2013 Nov 1;7(6):1461-9. doi: 10.1177/193229681300700606. PMID 24351172
- [Background] Jacobs PG, El Youssef J, Castle JR, Engle JM, Branigan DL, Johnson P, Massoud R, Kamath A, Ward WK. Development of a fully automated closed loop artificial pancreas control system with dual pump delivery of insulin and glucagon. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:397-400. doi: 10.1109/IEMBS.2011.6090127. PMID 22254332
- [Derived] Nguyen TP, Jacobs PG, Castle JR, Wilson LM, Kuehl K, Branigan D, Gabo V, Guillot F, Riddell MC, Haidar A, El Youssef J. Separating insulin-mediated and non-insulin-mediated glucose uptake during and after aerobic exercise in type 1 diabetes. Am J Physiol Endocrinol Metab. 2021 Mar 1;320(3):E425-E437. doi: 10.1152/ajpendo.00534.2020. Epub 2020 Dec 28. PMID 33356994